CLINICAL TRIAL: NCT03713112
Title: Efficacy and Feasibility of De-prescribing Rounds in a Singapore Rehabilitative Hospital- a Pilot Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bright Vision Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIRB Ref 2018/2721
Record Dates: First submitted 2018-10-12; First posted 2018-10-19 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Deprescribing; Multi-disciplinary; Rounds
Keywords: deprescribe; multi-disciplinary; open label; rounds; randomised controlled trial

STUDY DESIGN:
Intervention Model Description: The 2 arms of rehabilitative and/or subacute care patients consist of the intervention arm (receiving weekly multidisciplinary rounds up to the point of discharge, using 5 steps of deprescribing at the bedside, targeted to deprescribe selected medications [Beers' List of inappropriate Medications 2015; selected supplements and selected symptomatic medications]) and control arm (receving usual care)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekly MDT deprescribing rounds (Active Comparator): Weekly MDT deprescribing rounds for certain drugs will be performed on top of usual care.
  Interventions: Other: Weekly MDT deprescribing rounds for certain drugs
- Control (Usual Care) (No Intervention): Usual Care includes the following:
  * De-prescribing at the discretion of the ward doctors
  * Initial medication reconciliation by pharmacist on admission
  * Ward rounds to be conducted 3 weekdays per week for rehabilitative patients and daily on weekdays for sub-acute patients.

INTERVENTIONS:
Other: Weekly MDT deprescribing rounds for certain drugs — * Weekly deprescribing round (from randomization to day of discharge)
  * Conducted by a multidisciplinary team (non-ward doctors, pharmacist, ward nurse)
  * Using the 5 steps of de-prescribing
  * De-prescribing targets:
    1. Beer's list of potentially inappropriate medications (American Geriatric Society 2015 version)
    2. Supplements of questionable benefits (glucosamine, chondroitin, vitamin B complex and multivitamins)
    3. Symptomatic medications (laxatives, gastro-protectives, painkillers, anti-emetics and steroid creams) (Standardized verbal script to initiate de-prescribing by the team)
  * On top of usual care
  Arms: Weekly MDT deprescribing rounds

SUMMARY:
This open-labelled randomized control trial will be conducted in a Singapore Rehabilitation Hospital to investigate the efficacy, cost-reduction, safety and feasibility of a weekly deprescribing multi-disciplinary inpatient deprescribing round up to 28 days post discharge.

DETAILED DESCRIPTION:
ABSTRACT BACKGROUND: Deprescribing has been effective and safe in reducing polypharmacy and morbidity (e.g. fall), especially amongst elderly. However, little has been studied about the efficacy of a regular multidisciplinary round in deprescribing predefined medications in Singapore rehabilitative hospitals.

AIM: This study aims to evaluating the effects of a weekly multidisciplinary team(MDT) de-prescribing round on the reduction on total daily dose, cost of medications, its safety and feasibility in a Singapore rehabilitative hospital.

Methods: A total of 260 newly admitted patients will be randomised to a de-prescribing intervention (n= 130) or control (usual care) group (n= 130), using GraphPad randomization sequence software ©2017. The 5 steps of deprescribing process will be used and the targets of deprescribing are Beer's list of potentially inappropriate medications (AGS 2015 version), predetermined supplements and symptomatic medications. Predetermined medications were deprescribed following initial MDT assessment, discussion with attending doctors and consideration of patients' preferences regarding discontinuation or dose reduction. Total daily dose reduction, cost and side effects of deprescribing were monitored on admission day 14, 28, discharge day and post-discharge day 28. Time required for such rounds are also measured.

IMPACT: Once proven successful, this effective model of deprescribing could safely help to cut down caregiver's medicine administrative burden, improve compliance and reduce national healthcare cost. This model could also be easily replicated in all Singapore rehabilitative hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Greater or equals to 65 years old
* Newly admitted to rehabilitation or sub-acute disciplines
* Possess 1 or more of the targeted medications

Exclusion Criteria:

* Abbreviated mental test less than 7
* No mental capacity

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in total daily dose of medication upon discharge from the hospital | During the patient's inpatient stay (this will be measured on the day of discharge, usually ranging between 21 to 49 days upon inpatient admission)
  Change in total daily dose of medication upon discharge from the hospital

SECONDARY OUTCOMES:
Cost savings measured in Singapore dollars | These outcomes will be measured on days 14, 28 of inpatient admission, the day of inpatient discharge (*this is usually between 21 to 49 days after admission) and day 28 post discharge. Overall timeframe ranges between 49 to 77days after admission.
  Cost savings measured in Singapore dollars
Number of participants with side effects from deprescribing | These outcomes will be measured on days 14, 28 of inpatient admission, the day of inpatient discharge (*this is usually between 21 to 49 days after admission) and day 28 post discharge. Overall timeframe ranges between 49 to 77days after admission.
  Number of participants with side effects from deprescribing (i.e. recurrence of medical indications or symptoms; withdrawal effects of deprescribing; reinstating the same medications or substituting another medication, hospitalization and death)
feasibility of intervention in terms of time taken, measured in minutes. | During the patient's inpatient stay (this will be measured on the day of discharge, usually ranging between 21 to 49 days upon inpatient admission)
  The feasibility of implementation of intervention will also be determined through the time required to complete the de-prescribing process, measured in minutes.
feasibility of intervention in terms of ease at which the rounds are conducted (descriptive) | During the patient's inpatient stay (this will be measured on the day of discharge, usually ranging between 21 to 49 days upon inpatient admission)
  The feasibility of implementation of intervention will also be determined through limitations and challenges encountered, as documented by the multidisciplinary team.

CONTACTS AND LOCATIONS:
Overall Officials: Wong Peng Yong, Andrew, MBBS, Principal Investigator — Bright Vision Hospital; Singhealth Community Hospitals
Locations (1):
- Bright Vision Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
there's no current plans.

REFERENCES:
- [Result] Roberts MS, Stokes JA, King MA, Lynne TA, Purdie DM, Glasziou PP, Wilson DA, McCarthy ST, Brooks GE, de Looze FJ, Del Mar CB. Outcomes of a randomized controlled trial of a clinical pharmacy intervention in 52 nursing homes. Br J Clin Pharmacol. 2001 Mar;51(3):257-65. doi: 10.1046/j.1365-2125.2001.00347.x. PMID 11298072
- [Result] Kutner JS, Blatchford PJ, Taylor DH Jr, Ritchie CS, Bull JH, Fairclough DL, Hanson LC, LeBlanc TW, Samsa GP, Wolf S, Aziz NM, Currow DC, Ferrell B, Wagner-Johnston N, Zafar SY, Cleary JF, Dev S, Goode PS, Kamal AH, Kassner C, Kvale EA, McCallum JG, Ogunseitan AB, Pantilat SZ, Portenoy RK, Prince-Paul M, Sloan JA, Swetz KM, Von Gunten CF, Abernethy AP. Safety and benefit of discontinuing statin therapy in the setting of advanced, life-limiting illness: a randomized clinical trial. JAMA Intern Med. 2015 May;175(5):691-700. doi: 10.1001/jamainternmed.2015.0289. PMID 25798575
- [Result] Williams ME, Pulliam CC, Hunter R, Johnson TM, Owens JE, Kincaid J, Porter C, Koch G. The short-term effect of interdisciplinary medication review on function and cost in ambulatory elderly people. J Am Geriatr Soc. 2004 Jan;52(1):93-8. doi: 10.1111/j.1532-5415.2004.52016.x. PMID 14687321
- [Result] Reeve E, Andrews JM, Wiese MD, Hendrix I, Roberts MS, Shakib S. Feasibility of a patient-centered deprescribing process to reduce inappropriate use of proton pump inhibitors. Ann Pharmacother. 2015 Jan;49(1):29-38. doi: 10.1177/1060028014558290. Epub 2014 Nov 10. PMID 25385826
- [Result] Frank C, Weir E. Deprescribing for older patients. CMAJ. 2014 Dec 9;186(18):1369-76. doi: 10.1503/cmaj.131873. Epub 2014 Sep 2. No abstract available. PMID 25183716
- [Derived] Wong APY, Ting TW, Charissa EJM, Boon TW, Heng KY, Leng LL. Feasibility & Efficacy of Deprescribing rounds in a Singapore rehabilitative hospital- a randomised controlled trial. BMC Geriatr. 2021 Oct 21;21(1):584. doi: 10.1186/s12877-021-02507-0. PMID 34674645